CLINICAL TRIAL: NCT02429973
Title: Multicenter and Prospective Phase II Trial With Gemcitabine and Rapamycin in Second Line of Metastatic Osteosarcoma
Brief Title: Trial With Gemcitabine and Rapamycin in Second Line of Metastatic Osteosarcoma
Acronym: GEIS-29
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Broto, Javier Martín, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC11-444 OSTEOSARC
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Gemcitabine; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): 6 cycles of gemcitabine plus rapamycin
  Interventions: Drug: Gemcitabine plus rapamycin

INTERVENTIONS:
Drug: Gemcitabine plus rapamycin — Gemcitabine and rapamycin given in combination

SUMMARY:
Multicenter and prospective phase II trial with gemcitabine and rapamycin in second line of metastatic osteosarcoma. The study includes 6 cycles of the combination gemcitabine+rapamycin in metastatic or unresectable osteosarcoma patients.

DETAILED DESCRIPTION:
The trial seeks to analyze progression free survival (PFS), measured as PFS rate at 4 months, in patients with metastatic osteosarcoma who have previously received the most active drugs in this disease (methotrexate, cisplatin, adriamycin and ifosfamide). The treatment schedule consists of a maximum of 6 cycles of 3 weeks of gemcitabine+rapamycin. Gemcitabine is given at 800 mg/m2 in days 1 and 8 in cycles of 21 days. Rapamycin is given at 5 mg per day during treatment duration.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed before any trial test
* Age equal or less than 80 years
* Histological diagnosis of high-grade, metastatic or unresectable osteosarcoma in progression
* Previous treatment with drugs used in first line: methotrexate, adriamycin, platinum
* Measurable disease, acoording to RECIST criteria
* ECOG 0-2

Exclusion Criteria:

* Patients who have been irradiated on target lesions
* ECOG >2
* Bilirubin levels over normal values. Creatinine over 1.6 mg/dL
* History of other cancers except basal cell cancer or cervical cancer adequately treated
* Serious cardiovascular disease

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) rate | 4 months

SECONDARY OUTCOMES:
Tumor response according to RECIST | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martin, PhD, Principal Investigator — Virgen del Rocío Hospital